CLINICAL TRIAL: NCT01949987
Title: The Effect of Oral Intake on Pain Score in Children Undergoing Herniorrhaphy
Brief Title: Does Oral Intake Decreases Postoperative Pain Score in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibaraki Children's Hospital (Other)
Responsible Party: Principal Investigator, Kazuhiko Okuyama, MD, Chief anesthesiologist, Ibaraki Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pain and oral intake
Record Dates: First submitted 2013-09-09; First posted 2013-09-25 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Fasting; Postoperative Pain
MeSH Terms: conditions — Fasting; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 hours after surgery (Active Comparator): the investigators permit the patients to resume oral intake two hours after surgery and observe child's behavior and score; cry, facial expression, verbal expression, torso, legs, activity, and consolability
  Interventions: Other: two hours
- 1 hour after surgery (Experimental): the investigators permit the patients to resume oral intake one hour after surgery and observe child's behavior and score; cry, facial expression, verbal expression, torso, legs, activity, and consolability
  Interventions: Other: one hour

INTERVENTIONS:
Other: two hours
  Arms: 2 hours after surgery
Other: one hour
  Arms: 1 hour after surgery

SUMMARY:
Pain score after inguinal hernia repair surgery in children decreased as time passed in previous studies. Postoperative oral intake is usually resumed two hours after minor surgery in most of institutions, that may influence children's behavior and pain score.

A recent study suggest that oral intake one hour after minor surgery does not increase the incidence of postoperative nausea and vomiting.

The investigators primary endpoint is to clarify whether postoperative oral intake influences postoperative pain score in children.

ELIGIBILITY:
Inclusion Criteria:

* 18 month to 12 years old children undergoing elective unilateral inguinal hernia repair surgery

Exclusion Criteria:

* neurological disease, developmental delay

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
whether oral intake influences postoperative pain score in children | 90 minutes after surgery
  pain degree is assessed using mCHEOPS and FLACC in young children, and using FPS-R in older (8 years or older) children

SECONDARY OUTCOMES:
postoperative nausea and vomiting | 4 hours on average
  all children have to stay in hospital for 3 hours, and then, doctors visit the child and decide to discharge or not. Therefore, most of children stay in hospital approximately for 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiko Okuyama, MD, Study Director — Ibaraki Children's Hospital
Locations (1):
- Ibaraki Children's Hospital, Mito, Ibaraki, Japan